CLINICAL TRIAL: NCT00489528
Title: A Randomized, Parallel Group, Double-Blind, Placebo-Controlled, Dose-Ranging, Multicenter Study of Recombinant Human Growth Hormone (Serostim) in the Treatment of HIV-Associated Catabolism/Wasting
Brief Title: Growth Hormone in the Treatment of HIV-Associated Wasting
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: EMD Serono (Industry)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 9037; NCT00013988 (obsolete NCT alias)
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Last update posted 2013-10-22 (Estimated); Status verified 2013-10

CONDITIONS: HIV Infections; HIV Wasting Syndrome
Keywords: serostim; Dose-Response Relationship, Drug; Body Composition
MeSH Terms: conditions — HIV Infections; HIV Wasting Syndrome | interventions — Human Growth Hormone; Growth Hormone

INTERVENTIONS:
Drug: Somatropin; Recombinant human growth hormone (r hGH)

SUMMARY:
The purpose of this study is to compare physical function and lean body mass in patients getting different doses of somatropin compared to patients not getting the drug.

ELIGIBILITY:
Inclusion Criteria:

1. Have clearly documented HIV infection, determined by the presence of HIV confirmed by one of the following: Western blot, immunofluorescence assay, HIV culture, polymerase chain reaction (PCR) amplification, branched DNA (bDNA) signal amplification or the presence of p24 antigen. These tests may have been performed at any time in the past, but the results must be available for review by Serono prior to entry into the study.
2. Have evidence of AIDS wasting, with at least one of the following:

   * Documented unintentional weight loss of at least 10%, or
   * In the absence of unintentional weight loss of 10%, weight less than 90% of ideal body weight (Metropolitan Height and Weight Tables), or
   * In the absence of unintentional weight loss of 10%, body mass index < 20 kg/m².
3. Be at least 18 years of age.
4. Be receiving at least 90% of estimated caloric requirement on current nutritional regimen, according to a formal nutritional analysis.
5. Meet the following laboratory testing criteria at the week -4 visit (pre study screening):

   * AST, ALT, and amylase < 3 times the upper limit of normal.
   * Fasting triglyceride level < 500 mg/dl (or <5.64 mmol/l).
   * Fasting glucose < 110 mg/dl (or < 6.1mmol/l).
6. Be taking an antiretroviral medication that is approved or available under a Treatment IND (in the US) or a temporary approval (outside the US).

   * The subject must have been on the antiretroviral therapy for at least 8 weeks prior to study Day 1.
   * The subject must agree not to change the antiviral regimen during the 12 weeks of study drug administration (unless medically mandated).
7. Be capable of completing all required study activities and assessments (including all required exercise performance tests).
8. Understand and sign an informed consent document.

Exclusion Criteria:

1. Any medical history of the following:

   * Pancreatitis.
   * Carpal tunnel syndrome (unless resolved by surgical release).
   * Glucose intolerance [for the purpose of this protocol defined as fasting blood glucose ≥ 110 mg/dl (6.1 mmol/l), or 2 hour/random blood glucose ≥ 140 mg/dl (7.8 mg/dl)].
   * Angina pectoris.
   * Coronary artery disease.
   * Any disorder associated with moderate to severe edema (e.g., cirrhosis, nephrosis, congestive heart failure, lymphedema).
   * Allergy or hypersensitivity to growth hormone.
2. Any of the following medical conditions:

   * Active AIDS-defining opportunistic infection.
   * Any active malignancy, except for localized cutaneous Kaposi's sarcoma (fewer than 10 lesions, none of which exceeds 2 cm in size, not on active therapy).
   * A central nervous system (CNS) mass, or CNS process associated with active neurological findings.
   * Chronic diarrhea (defined as 6 or more liquid stools per day).
   * Unstable or untreated hypertension.
3. Patients with acute critical illnesses in intensive care units due to complications following open heart or abdominal surgery, multiple accidental trauma, or with acute respiratory failure.
4. Either of the following aspects of the medical regimen in the 30 days prior to study entry (60 days prior to receiving study drug):

   * New systemic therapy for opportunistic infection.
   * New therapy for wasting, including parenteral or oral hyperalimentation, tube feeding, anabolic or progestational agents, or appetite stimulants.
5. Prior radiation therapy or systemic chemotherapy.
6. Use of glucocorticoids within the past six months or growth hormone within the past year.
7. An untreated or suspected serious systemic infection, or persistent fever > 101°F (or 38.5°C) during the 30 days prior to study entry.
8. Evidence of gastrointestinal (GI) bleeding, obstruction, or malabsorption as determined by the Investigator.
9. Active substance abuse which would prevent informed consent or compliance with study activities.
10. Dementia which would preclude the patient from giving informed consent or complying with the requirements of this protocol.
11. If female, be neither pregnant or breast feeding.
12. Use of an investigational agent under another protocol unless discussed and approved in advance by Serono's Therapeutic Director.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 1997-07; Study Completion 2002-03 (Actual)

PRIMARY OUTCOMES:
To confirm the clinical efficacy of Serostim compared with placebo, based on an endpoint of exercise function change.

SECONDARY OUTCOMES:
To establish an optimal dose of Serostim, based on the endpoint of lean body mass (LBM) change.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth Svanbert, MD, PhD, Study Director